CLINICAL TRIAL: NCT02738151
Title: A 24-week, Multicenter, Randomized, Open-Label, Parallel-group StudyComparing the Efficacy and Safety of Toujeo® and Tresiba® in Insulin-NaivePatients With Type 2 Diabetes Mellitus Not Adequately Controlled With OralAntihyperglycemic Drug(s) ± GLP-1 Receptor Agonist
Brief Title: Efficacy and Safety of Toujeo® Versus Tresiba® in Insulin-Naive Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Oral Antihyperglycemic Drug(s) ± GLP-1 Receptor Agonist
Acronym: BRIGHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS14584; 2015-005101-36 (EudraCT Number); U1111-1177-6327 (Other: UTN)
Record Dates: First submitted 2016-03-31; First posted 2016-04-14 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toujeo (Experimental): Toujeo® (Insulin glargine, 300 U/mL) subcutaneous (SC) injection once daily up to Week 24 on top of non-insulin antidiabetic treatment.
  Interventions: Drug: Insulin glargine, 300U/mL; Drug: Non-insulin anti-diabetic treatment
- Tresiba (Active Comparator): Tresiba® (Insulin Degludec, 100 U/mL) SC injection once daily up to Week 24 on top of non-insulin antidiabetic treatment .
  Interventions: Drug: Insulin degludec, 100 U/mL; Drug: Non-insulin anti-diabetic treatment

INTERVENTIONS:
Drug: Insulin glargine, 300U/mL — Self-administered by subcutaneous (SC) injection in the evening using a pre-filled pen. Dose titration to achieve fasting self-monitored plasma glucose (SMPG) from 80 to 100 mg/dL (4.4 to 5.6 mmol/L).
  Other Names: HOE901-U300; Toujeo
  Arms: Toujeo
Drug: Insulin degludec, 100 U/mL — Self-administered by subcutaneous (SC) injection in the evening using a pre-filled pen. Dose titration to achieve fasting self-monitored plasma glucose (SMPG) from 80 to 100 mg/dL (4.4 to 5.6 mmol/L).
  Route of administration: subcutaneous
  Other Names: Tresiba
  Arms: Tresiba
Drug: Non-insulin anti-diabetic treatment — Background therapy: Oral Anti diabetics Drugs (OADs), Glucagon-like peptide-1 (GLP-1) receptor agonist.

SUMMARY:
Primary Objective:

To demonstrate the noninferiority in the efficacy of Toujeo® to Tresiba® in glycated hemoglobin (HbA1c) change from Baseline to Week 24.

Secondary Objectives:

Change From Baseline in HbA1c to Week 12

To assess the effects of the insulin Toujeo® in comparison with insulin Tresiba® at week 12 and week 24 on:

* Change in Fasting plasma glucose (FPG);
* Change in Fasting self-monitored plasma glucose (SMPG) and 4-point SMPG and 8-point SMPG profile;
* Percentage of participants reaching HbA1c targets <7% or ≤6.5%;
* Percentage of participants reaching HbA1c targets <7% or ≤6.5% without severe and/or confirmed hypoglycemia
* Frequency of occurrence and diurnal distribution of hypoglycemia by American Diabetes Association (ADA) category of hypoglycemia.

To assess the safety in each treatment group.

To assess the treatment effects in each treatment group on Patient Reported Outcomes (PRO).

Percentage of participants requiring rescue therapy.

DETAILED DESCRIPTION:
The maximum study duration per participant was approximately 27 weeks: an up to 2-week screening period, a 24-week randomized treatment period (including 12 weeks active titration), and a 7-day posttreatment safety follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Adult participants with type 2 diabetes mellitus (T2DM) inadequately controlled with OADs therapy with/without GLP-1 receptor agonist at stable dose for at least 3 months.
* Signed written informed consent.

Exclusion criteria:

* Age <18 years.
* HbA1c <7.5% or >10.5% (at screening visit). Body mass index (BMI) <25 kg/m^2 or >40 kg/m^2.
* History of T2DM for less than 1 year before screening.
* Less than 6 months before screening on OADs treatment and GLP-1 receptor agonist (if taken).
* Current or previous insulin use except for a maximum of 8 consecutive days or totally 15 days (eg, acute illness, surgery) during the last year prior to screening.
* Initiation of new glucose-lowering medications and/or weight loss drug in the last 3 months before screening visit.
* Participant receiving only noninsulin antihyperglycemic drugs not approved for combination with insulin according to local labelling/local treatment guideline.
* History of hypoglycemia unawareness or repeated episodes of severe hypoglycemia or metabolic acidosis, including hospitalization for diabetic ketoacidosis during the last 12 months prior to screening.
* Unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to require treatment (eg, laser, surgical treatment, or injectable drugs) during the study period.
* End stage renal disease.
* Any acute or chronic condition that in the opinion of Investigator would affect the safety of participant, compliance, or study results.
* Any contraindication to use of Toujeo® or Tresiba® as defined in the national product label, hypersensitivity to Toujeo® or Tresiba® active ingredients or one of the excipients.
* Pregnant or breast-feeding women.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 929 (Actual)
Dates: Start 2016-05-19; Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (158):
- United States (74):
  - Investigational Site Number 840038, Sheffield, Alabama
  - Investigational Site Number 840066, Phoenix, Arizona
  - Investigational Site Number 840051, Anaheim, California
  - Investigational Site Number 840081, Chino, California
  - Investigational Site Number 840016, Huntington Park, California
  - Investigational Site Number 840002, La Jolla, California
  - Investigational Site Number 840091, Los Angeles, California
  - Investigational Site Number 840058, Northridge, California
  - Investigational Site Number 840021, Palm Springs, California
  - Investigational Site Number 840087, Santa Ana, California
  - Investigational Site Number 840030, Torrance, California
  - Investigational Site Number 840065, Van Nuys, California
  - Investigational Site Number 840075, Bradenton, Florida
  - Investigational Site Number 840076, New Port Richey, Florida
  - Investigational Site Number 840026, Ocoee, Florida
  - Investigational Site Number 840052, Palm Harbor, Florida
  - Investigational Site Number 840080, Palm Harbor, Florida
  - Investigational Site Number 840018, Port Charlotte, Florida
  - Investigational Site Number 840071, Lawrenceville, Georgia
  - Investigational Site Number 840085, Roswell, Georgia
  - Investigational Site Number 840072, Statesboro, Georgia
  - Investigational Site Number 840039, Stockbridge, Georgia
  - Investigational Site Number 840036, Arlington Heights, Illinois
  - Investigational Site Number 840010, Chicago, Illinois
  - Investigational Site Number 840005, Avon, Indiana
  - Investigational Site Number 840063, Council Bluffs, Iowa
  - Investigational Site Number 840098, Des Moines, Iowa
  - Investigational Site Number 840101, Des Moines, Iowa
  - Investigational Site Number 840096, West Des Moines, Iowa
  - Investigational Site Number 840061, Paris, Kentucky
  - Investigational Site Number 840011, Hyattsville, Maryland
  - Investigational Site Number 840001, Rockville, Maryland
  - Investigational Site Number 840041, Flint, Michigan
  - Investigational Site Number 840057, Flint, Michigan
  - Investigational Site Number 840033, Troy, Michigan
  - Investigational Site Number 840084, Olive Branch, Mississippi
  - Investigational Site Number 840048, Chesterfield, Missouri
  - Investigational Site Number 840023, Las Vegas, Nevada
  - Investigational Site Number 840045, Las Vegas, Nevada
  - Investigational Site Number 840031, Linden, New Jersey
  - Investigational Site Number 840060, Hickory, North Carolina
  - Investigational Site Number 840064, Morganton, North Carolina
  - Investigational Site Number 840043, Wilmington, North Carolina
  - Investigational Site Number 840082, Winston-Salem, North Carolina
  - Investigational Site Number 840025, Oklahoma City, Oklahoma
  - Investigational Site Number 840022, Oklahoma City, Oklahoma
  - Investigational Site Number 840029, Beaver, Pennsylvania
  - Investigational Site Number 840056, Downingtown, Pennsylvania
  - Investigational Site Number 840093, Anderson, South Carolina
  - Investigational Site Number 840097, Greenville, South Carolina
  - Investigational Site Number 840070, Greer, South Carolina
  - Investigational Site Number 840044, North Myrtle Beach, South Carolina
  - Investigational Site Number 840069, Simpsonville, South Carolina
  - Investigational Site Number 840079, Bristol, Tennessee
  - Investigational Site Number 840006, Chattanooga, Tennessee
  - Investigational Site Number 840088, Knoxville, Tennessee
  - Investigational Site Number 840077, New Tazewell, Tennessee
  - Investigational Site Number 840007, Dallas, Texas
  - Investigational Site Number 840086, Dallas, Texas
  - Investigational Site Number 840027, Houston, Texas
  - Investigational Site Number 840004, Houston, Texas
  - Investigational Site Number 840040, Houston, Texas
  - Investigational Site Number 840046, Houston, Texas
  - Investigational Site Number 840054, Hurst, Texas
  - Investigational Site Number 840017, Mesquite, Texas
  - Investigational Site Number 840008, Missouri City, Texas
  - Investigational Site Number 840094, San Antonio, Texas
  - Investigational Site Number 840009, Sugar Land, Texas
  - Investigational Site Number 840053, Waco, Texas
  - Investigational Site Number 840095, Ogden, Utah
  - Investigational Site Number 840032, Salt Lake City, Utah
  - Investigational Site Number 840024, Norfolk, Virginia
  - Investigational Site Number 840020, Richmond, Virginia
  - Investigational Site Number 840012, Renton, Washington
- Bulgaria (3):
  - Investigational Site Number 100001, Sofia
  - Investigational Site Number 100002, Sofia
  - Investigational Site Number 100003, Sofia
- Croatia (3):
  - Investigational Site Number 191001, Rijeka
  - Investigational Site Number 191002, Rijeka
  - Investigational Site Number 191003, Zagreb
- Czechia (8):
  - Investigational Site Number 203009, Hlučín
  - Investigational Site Number 203006, Jílové u Prahy
  - Investigational Site Number 203005, Liberec
  - Investigational Site Number 203001, Pardubice
  - Investigational Site Number 203007, Prague
  - Investigational Site Number 203008, Prague
  - Investigational Site Number 203002, Prague
  - Investigational Site Number 203004, Vsetín
- Denmark (4):
  - Investigational Site Number 208003, Aarhus
  - Investigational Site Number 208002, Hillerød
  - Investigational Site Number 208001, København NV
  - Investigational Site Number 208004, Odense
- France (6):
  - Investigational Site Number 250002, La Roche-sur-Yon
  - Investigational Site Number 250003, La Rochelle
  - Investigational Site Number 250001, Nantes
  - Investigational Site Number 250006, Nîmes
  - Investigational Site Number 250005, Poitiers
  - Investigational Site Number 250007, Vénissieux
- Greece (4):
  - Investigational Site Number 300005, Alexandroupoli
  - Investigational Site Number 300001, Athens
  - Investigational Site Number 300002, Athens
  - Investigational Site Number 300003, Athens
- Hungary (4):
  - Investigational Site Number 348004, Budapest
  - Investigational Site Number 348002, Budapest
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348003, Gyöngyös
- Israel (8):
  - Investigational Site Number 376001, Haifa
  - Investigational Site Number 376004, Haifa
  - Investigational Site Number 376008, Haifa
  - Investigational Site Number 376009, Kfar Saba
  - Investigational Site Number 376002, Petah Tikva
  - Investigational Site Number 376006, Tel Aviv
  - Investigational Site Number 376007, Tel Aviv
  - Investigational Site Number 376003, Tel Litwinsky
- Italy (12):
  - Investigational Site Number 380007, Bari
  - Investigational Site Number 380009, Catanzaro
  - Investigational Site Number 380010, Chieti
  - Investigational Site Number 380014, Milan
  - Investigational Site Number 380002, Moncalieri
  - Investigational Site Number 380011, Napoli
  - Investigational Site Number 380008, Roma
  - Investigational Site Number 380015, Roma
  - Investigational Site Number 380016, Roma
  - Investigational Site Number 380013, Sesto San Giovanni
  - Investigational Site Number 380005, Torino
  - Investigational Site Number 380012, Verona
- Romania (13):
  - Investigational Site Number 642007, Brasov
  - Investigational Site Number 642008, Brasov
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642013, Bucharest
  - Investigational Site Number 642015, Bucharest
  - Investigational Site Number 642003, Cluj-Napoca
  - Investigational Site Number 642009, Constanța
  - Investigational Site Number 642014, Iași
  - Investigational Site Number 642005, Oradea
  - Investigational Site Number 642012, Oradea
  - Investigational Site Number 642010, Târgu Mureş
  - Investigational Site Number 642004, Târgu Mureş
  - Investigational Site Number 642006, Târgu Mureş
- Serbia (3):
  - Investigational Site Number 688001, Belgrade
  - Investigational Site Number 688002, Niš
  - Investigational Site Number 688003, Niš
- Slovakia (5):
  - Investigational Site Number 703006, Košice
  - Investigational Site Number 703002, Ľubochňa
  - Investigational Site Number 703001, Moldava nad Bodvou
  - Investigational Site Number 703003, Sabinov
  - Investigational Site Number 703005, Trebišov
- Sweden (2):
  - Investigational Site Number 752102, Lund
  - Investigational Site Number 752101, Skövde
- Switzerland (2):
  - Investigational Site Number 756003, Olten
  - Investigational Site Number 756001, Sankt Gallen
- United Kingdom (7):
  - Investigational Site Number 826001, Chertsey
  - Investigational Site Number 826005, Gillingham
  - Investigational Site Number 826008, Lincoln
  - Investigational Site Number 826002, London
  - Investigational Site Number 826009, Manchester
  - Investigational Site Number 826006, Margate
  - Investigational Site Number 826004, Swansea

REFERENCES:
- [Derived] Rosenstock J, Cheng A, Ritzel R, Bosnyak Z, Devisme C, Cali AMG, Sieber J, Stella P, Wang X, Frias JP, Roussel R, Bolli GB. More Similarities Than Differences Testing Insulin Glargine 300 Units/mL Versus Insulin Degludec 100 Units/mL in Insulin-Naive Type 2 Diabetes: The Randomized Head-to-Head BRIGHT Trial. Diabetes Care. 2018 Oct;41(10):2147-2154. doi: 10.2337/dc18-0559. Epub 2018 Aug 13. PMID 30104294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 158 study centers across 16 countries. A total of 1376 participants were screened between 19 May 2016 and 19 February 2017, of whom 447 were screen failures.
Pre-assignment Details: A total of 929 participants were randomized in 1:1 ratio to either Toujeo or Tresiba, stratified by screening glycated hemoglobin (HbA1c) values (<8% or >=8%); and use of sulfonylurea (SU) or meglitinides before the day of screening ('yes' versus 'no').
Groups:
- Tresiba: Tresiba® (Insulin Degludec, 100 U/mL) SC injection once daily up to Week 24 on top of non-insulin antidiabetic treatment.
Period: Overall Study
Arm/Group | Toujeo | Tresiba
Started | 466 | 463
Treated | 462 | 462
Completed | 443 | 432
Not Completed | 23 | 31
Not completed — Randomized but not treated | 4 | 1
Not completed — Adverse Event | 4 | 5
Not completed — Hypoglycemia | 0 | 1
Not completed — Poor Compliance to Protocol | 4 | 3
Not completed — Other than specified above | 11 | 21

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Toujeo: Toujeo® (Insulin glargine, 300 U/mL) SC injection once daily up to Week 24 on top of non-insulin antidiabetic treatment.
- Total: Total of all reporting groups
Arm/Group | Toujeo | Tresiba | Total
Number analyzed (Participants) | 466 | 463 | 929
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.6) | 60.5 (9.8) | 60.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 219 | 211 | 430
  Male | 247 | 252 | 499
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 31.7 (4.3) | 31.3 (4.4) | 31.5 (4.4)
Duration of Type 2 Diabetes Mellitus [Mean (Standard Deviation); unit: years] | 10.5 (6.1) | 10.7 (6.5) | 10.6 (6.3)
Baseline HbA1c [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.71 (0.83) | 8.57 (0.80) | 8.64 (0.82)
Basal Insulin Daily Dose [Mean (Standard Deviation); unit: Units per kilogram (U/kg)] — Population: Number of participants analyzed = participants with available data for specified measure.
  Units per kilogram (U/kg)
    number analyzed (Participants) | 461 | 461 | 922
    (all) | 0.19 (0.04) | 0.12 (0.03) | 0.15 (0.05)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c to Week 24
Description: Change in HbA1c was calculated by subtracting baseline value from Week 24 value. Adjusted Least Square (LS) means and standard errors were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data, using all post-baseline HbA1c data available during the 24-week on-treatment period.
Time Frame: Baseline, Week 24
Population: Intent-to-treat(ITT) population: all randomized participants who received at least 1 dose of IMP, regardless of whether treatment was actually being received & analyzed as per allocated treatment group. Overall number of participants analyzed=participants with at least 1 baseline & 1 post-baseline HbA1c assessment during 24week on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 430 | 425
percentage of HbA1c | -1.64 (0.037) | -1.59 (0.037)
Statistical Analysis 1: Comparison: Toujeo vs Tresiba; A hierarchical step-down testing procedure was used to control type 1 error. Analysis was performed using a MMRM approach with treatment groups, randomization strata, visit, and treatment-by-visit interaction as fixed categorical effects and baseline HbA1c value and baseline HbA1c value-by-visit interaction as continuous fixed covariates; Test type: Non-Inferiority — Non-inferiority of Toujeo vs Tresiba was demonstrated if the upper bound of the two-sided 95% confidence interval (CI) for the difference between groups was <0.3%; p < .0001, Mixed Models Analysis — Threshold for significance at 0.025 level; Least Square (LS) Mean difference = -0.05, 95% CI 2-sided [-0.152 to 0.051], Standard Error of Mean 0.052 — Toujeo vs. Tresiba
Statistical Analysis 2: Comparison: Toujeo vs Tresiba; Superiority of Toujeo over Tresiba was demonstrated if the upper bound of the two-sided 95% CI for the difference in the mean change in HbA1c from baseline to Week 24 between Toujeo over Tresiba on ITT population was <0 (zero); Test type: Superiority; p = 0.3302, Mixed Models Analysis; LS Mean Difference = -0.05, 95% CI 2-sided [-0.152 to 0.051], Standard Error of Mean 0.052

2. Secondary Outcome: Change From Baseline in HbA1c to Week 12
Description: Change in HbA1c was calculated by subtracting baseline value from Week 12 value. Adjusted least square means and standard errors were obtained from a mixed-effect model with MMRM.
Time Frame: Baseline, Week 12
Population: ITT population. Here, overall number of participants analyzed = participants with at least one baseline and one post-baseline HbA1c assessment during the 12 week on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 448 | 445
percentage of HbA1c | -1.37 (0.036) | -1.39 (0.036)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) to Week 12 and Week 24
Description: Change in FPG was calculated by subtracting baseline value from Week 12 and Week 24 value. Adjusted LS means were obtained from MMRM including post baseline values during the 24-week on-treatment period.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT population. Here, number analyzed = participants with at least one baseline and one post baseline FPG values at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
mmol/L
  Week 12: number analyzed (Participants) | 442 | 441
  Week 12 | -3.64 (0.099) | -3.89 (0.100)
  Week 24: number analyzed (Participants) | 417 | 408
  Week 24 | -3.52 (0.109) | -3.95 (0.110)

4. Secondary Outcome: Change From Baseline in Fasting Self-Monitoring Plasma Glucose (SMPG) to Week 12 and Week 24
Description: Fasting SMPG was measured by the participant before breakfast and before the administration of the glucose-lowering agents once a day during the study. Adjusted LS means were obtained from MMRM including post baseline values during the 24 week on treatment period.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT population. Here, overall number analyzed =participants with at least one baseline and one post baseline fasting SMPG values at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
mmol/L
  Week 12: number analyzed (Participants) | 430 | 431
  Week 12 | -3.26 (0.067) | -3.25 (0.067)
  Week 24: number analyzed (Participants) | 421 | 416
  Week 24 | -3.23 (0.067) | -3.29 (0.068)

5. Secondary Outcome: Change From Baseline in 8 Point SMPG Profile to Week 12 and Week 24 Per Time Point
Description: 8-point SMPG profiles were measured at the following 8 points: 03:00 at night, pre-breakfast, 2 hours after breakfast, pre-lunch, 2 hours after lunch, pre-dinner, 2 hours after dinner, and bedtime.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT population. Number Analyzed = participants with at least one baseline and one post baseline 8 Point SMPG values at specified time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
mmol/L
  Week 12: 03:00 at night: number analyzed (Participants) | 342 | 334
  Week 12: 03:00 at night | -2.77 (3.16) | -2.28 (3.49)
  Week 12: Pre-breakfast: number analyzed (Participants) | 378 | 371
  Week 12: Pre-breakfast | -3.42 (2.79) | -3.00 (2.63)
  Week 12: 2 hours after breakfast: number analyzed (Participants) | 365 | 351
  Week 12: 2 hours after breakfast | -3.20 (4.02) | -3.23 (3.92)
  Week 12: Pre-lunch: number analyzed (Participants) | 365 | 358
  Week 12: Pre-lunch | -2.64 (3.90) | -2.50 (3.65)
  Week 12: 2 hours after lunch: number analyzed (Participants) | 365 | 367
  Week 12: 2 hours after lunch | -2.51 (4.15) | -1.99 (3.94)
  Week 12: Pre-dinner: number analyzed (Participants) | 366 | 363
  Week 12: Pre-dinner | -2.04 (3.63) | -1.93 (3.74)
  Week 12: 2 hours after dinner: number analyzed (Participants) | 355 | 352
  Week 12: 2 hours after dinner | -2.32 (4.20) | -1.76 (3.87)
  Week 12: Bedtime: number analyzed (Participants) | 344 | 331
  Week 12: Bedtime | -2.44 (4.07) | -2.08 (3.95)
  Week 24: 03:00 at night: number analyzed (Participants) | 331 | 305
  Week 24: 03:00 at night | -2.65 (3.43) | -2.43 (3.51)
  Week 24: Pre-breakfast: number analyzed (Participants) | 363 | 341
  Week 24: Pre-breakfast | -3.37 (2.81) | -3.03 (2.85)
  Week 24: 2 hours after breakfast: number analyzed (Participants) | 346 | 326
  Week 24: 2 hours after breakfast | -3.30 (3.68) | -3.50 (4.00)
  Week 24: Pre-lunch: number analyzed (Participants) | 350 | 331
  Week 24: Pre-lunch | -2.81 (3.67) | -2.29 (3.93)
  Week 24: 2 hours after lunch: number analyzed (Participants) | 350 | 338
  Week 24: 2 hours after lunch | -2.74 (3.73) | -1.93 (3.91)
  Week 24: Pre-dinner: number analyzed (Participants) | 350 | 333
  Week 24: Pre-dinner | -1.87 (3.78) | -1.86 (4.01)
  Week 24: 2 hours after dinner: number analyzed (Participants) | 338 | 326
  Week 24: 2 hours after dinner | -2.28 (4.19) | -2.07 (4.00)
  Week 24: Bedtime: number analyzed (Participants) | 315 | 286
  Week 24: Bedtime | -2.52 (3.87) | -2.09 (3.96)

6. Secondary Outcome: Change From Baseline in 4-point SMPG Profile to Week 12 and Week 24 Per Time Point
Description: 4-point SMPG profiles were measured at the following 4 points: prebreakfast, prelunch, predinner and bedtime.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT population. Number analyzed = Participants with at least one baseline and one post-baseline 4-point SMPG values at specified timepoints.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
mmol/L
  Week 12: Pre-breakfast: number analyzed (Participants) | 380 | 374
  Week 12: Pre-breakfast | -3.41 (2.75) | -2.97 (2.62)
  Week 12: Pre-lunch: number analyzed (Participants) | 369 | 362
  Week 12: Pre-lunch | -2.63 (3.88) | -2.44 (3.65)
  Week 12: Pre-dinner: number analyzed (Participants) | 371 | 370
  Week 12: Pre-dinner | -2.03 (3.64) | -1.92 (3.76)
  Week 12: Bedtime: number analyzed (Participants) | 346 | 336
  Week 12: Bedtime | -2.41 (4.10) | -2.11 (3.96)
  Week 24: Pre-breakfast: number analyzed (Participants) | 363 | 341
  Week 24: Pre-breakfast | -3.38 (2.81) | -2.99 (2.81)
  Week 24: Pre-lunch: number analyzed (Participants) | 351 | 332
  Week 24: Pre-lunch | -2.81 (3.67) | -2.26 (3.92)
  Week 24: Pre-dinner: number analyzed (Participants) | 353 | 335
  Week 24: Pre-dinner | -1.88 (3.79) | -1.86 (4.01)
  Week 24: Bedtime: number analyzed (Participants) | 314 | 289
  Week 24: Bedtime | -2.51 (3.87) | -2.10 (4.00)

7. Secondary Outcome: Change From Baseline in 24-hour Average 8-point SMPG Profile to Week 12 and Week 24
Description: The 8-point SMPG profile was measured at the following 8 points: 03:00 at night, pre-breakfast, 2 hours after breakfast, pre-lunch, 2 hours after lunch, pre-dinner, 2 hours after dinner, and bedtime. Adjusted LS means were obtained from MMRM.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT population. Here, number analyzed = Participants with at least one baseline and one post-baseline 24-hour average SMPG values at specified time points.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
mmol/L
  Week 12: number analyzed (Participants) | 379 | 375
  Week 12 | -2.57 (0.092) | -2.50 (0.093)
  Week 24: number analyzed (Participants) | 363 | 345
  Week 24 | -2.62 (0.094) | -2.53 (0.096)

8. Secondary Outcome: Change From Baseline in Variability of Fasting SMPG to Week 12 and Week 24
Description: Adjusted LS means were obtained from MMRM. Variability was assessed by the mean of coefficient of variation calculated over at least 3 SMPG measured during the 7 days preceding the given visit.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT population. Number Analyzed = participants with at least one baseline and one post baseline Fasting SMPG values at specified time point.
Measure: Least Squares Mean (Standard Error); unit: percentage of mean variability
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
percentage of mean variability
  Week 12: number analyzed (Participants) | 430 | 431
  Week 12 | 2.38 (0.418) | 2.62 (0.416)
  Week 24: number analyzed (Participants) | 421 | 416
  Week 24 | 1.49 (0.391) | 1.97 (0.390)

9. Secondary Outcome: Change From Baseline in Variability of 24-Hour 8-Point SMPG Profiles at Week 12 and Week 24
Description: Adjusted LS means were obtained from MMRM.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: percentage of mean variability
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
percentage of mean variability
  Week 12: number analyzed (Participants) | 379 | 375
  Week 12 | 4.08 (0.562) | 4.73 (0.561)
  Week 24: number analyzed (Participants) | 363 | 345
  Week 24 | 3.70 (0.588) | 3.95 (0.599)

10. Secondary Outcome: Percentage of Participants Reaching Target HbA1c of < 7% and =<6.5% at Week 12 and Week 24
Description: Only the post-baseline HbA1c measurements before rescue and during the 12 week and 24-week on-treatment period were considered in the analysis.
Time Frame: Week 12, and Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
percentage of participants
  Participants who reached the target <7% at Week 12 | 34.63 | 36.15
  Participants who reached target <=6.5% at Week 12 | 11.47 | 14.29
  Participants who reached the target <7% at Week 24 | 48.70 | 44.59
  Participants who reached target <=6.5% at Week 24 | 21.21 | 19.70

11. Secondary Outcome: Percentage of Participants Reaching Target HbA1c <7% and =<6.5% at Week 12 and Week 24 Without Severe and/or Confirmed Hypoglycemia (70 mg/dL) Event
Description: Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Severe and/or confirmed hypoglycemia event was a severe event or an event confirmed by plasma glucose =<3.9 mmol/L (=<70 mg/dL).
Time Frame: Week 12, and Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
percentage of participants
  Week12: Participants who reached the target <7% | 16.45 | 13.64
  Week12: Participants who reached target <=6.5% | 4.11 | 4.55
  Week24: Participants who reached the target <7% | 13.42 | 12.99
  Week24: Participants who reached target <=6.5% | 5.84 | 5.19

12. Secondary Outcome: Percentage of Participants With Sulphonylurea or Meglitinide Dose Reduction/ Discontinuation Due to Hypoglycemia During 24 Weeks Treatment Period
Description: Percentage of participants With Sulphonylurea or Meglitinide dose reduction/ discontinuation due to Hypoglycemia during 24 Week treatment period were reported. Only participants with Sulphonylurea or meglitinides at Screening as per actual strata were taken into account in this analysis.
Time Frame: Baseline to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
percentage of participants | 4.98 | 4.76

13. Secondary Outcome: Percentage of Participants Requiring a Rescue Therapy During 24 Weeks Treatment Period
Description: Routine fasting SMPG and central laboratory FPG (and HbA1c after Week 12) values were used to determine the requirement of rescue medication. Threshold values at Week 12: FPG >200 mg/dL (11 mmol/L), or HbA1c >8.5%.
Time Frame: Baseline to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
percentage of participants | 1.30 | 1.30

14. Secondary Outcome: Change From Baseline in Basal Insulin Dose (U/kg Body Weight) to Week 12 and Week 24
Description: Only the insulin dose measurements performed before initiation of rescue therapy and during the on-treatment period were considered in the analysis.
Time Frame: Baseline, Week 12 and Week 24
Population: Safety population included all randomized participants who did actually receive at least one dose of IMP, regardless of the amount of treatment administered.
Measure: Mean (Standard Deviation); unit: Units per kilogram (U/kg)
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
Units per kilogram (U/kg)
  Week 12: number analyzed (Participants) | 450 | 445
  Week 12 | 0.289 (0.200) | 0.255 (0.195)
  Week 24: number analyzed (Participants) | 436 | 425
  Week 24 | 0.357 (0.253) | 0.309 (0.241)

15. Secondary Outcome: Percentage of Participants With At Least One Hypoglycemic Events (Any, Severe and/or Confirmed Hypoglycemia: Any Time of the Day) by Study Period
Description: Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Severe and/or confirmed hypoglycemia event was a severe event or an event confirmed with plasma glucose =<70 mg/dL (=<3.9 mmol/L), or < 54 mg/dL (<3.0 mmol/L). Assessment was done by treatment period (for =<12 weeks, for >12 weeks to =<24 weeks (24W)). Percentage of participants with at least one hypoglycemia (hypo) event at any time of the day were reported.
Time Frame: Day 1-Week 12, Week 13-Week 24, and 24 Week Period
Population: Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
percentage of participants
  Any hypo Day1-Week 12 | 53.0 | 58.4
  Any hypo Week13-14 | 57.2 | 57.4
  Any hypo 24 week period | 70.1 | 71.2
  Severe and/or confirmed hypo (=<70mg/dL) D1-W12 | 47.4 | 54.3
  Severe and/or confirmed hypo (=<70mg/dL) W13-14 | 54.1 | 55.8
  Severe and/or confirmed hypo(=<70mg/dL) 24W period | 66.5 | 69.0
  Severe and/or confirmed hypo (< 54mg/dL) D1-W12 | 7.8 | 11.7
  Severe and/or confirmed hypo( <54 mg/dL) W13-14 | 9.8 | 11.2
  Severe and/or confirmed hypo (<54mg/dL) 24W period | 14.7 | 18.4

16. Secondary Outcome: Percentage of Participants With At Least One Hypoglycemic Events (Any, Severe and/or Confirmed Hypoglycemia: Nocturnal) by Study Period
Description: Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Severe and/or confirmed hypoglycaemia event was a severe event or an event confirmed with plasma glucose =<70 mg/dL (=<3.9 mmol/L), or < 54 mg/dL (<3.0 mmol/L). Nocturnal hypoglycemia was hypoglycemia that occurred between 00:00 and 05:59 hours (clock time). Assessment was done by treatment period (for =<12 weeks, for >12 weeks to =<24 weeks).
Time Frame: Day 1-Week 12, Week 13-Week 24, and 24 Week Period
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
percentage of participants
  Any hypo D1-W12 | 18.4 | 21.0
  Any hypo W13-14 | 22.7 | 21.2
  Any hypo 24Week period | 31.2 | 30.3
  Severe and/or confirmed hypo (=<70mg/dL)D1-W12 | 15.2 | 18.8
  Severe and/or confirmed hypo (=<70mg/dL)W13-14 | 21.4 | 21.0
  Severe and/or confirmed hypo(=<70mg/dL)24W Period | 28.6 | 28.8
  Severe and/or confirmed hypo(< 54mg/dL)D1-W12 | 2.8 | 3.5
  Severe and/or confirmed hypo(< 54mg/dL)W13-14 | 4.5 | 3.8
  Severe and/or confirmed hypo(< 54mg/dL)24W Period | 6.1 | 6.1

17. Secondary Outcome: Hypoglycemia (Any, Severe and/or Confirmed Hypoglycemia: Any Time of the Day) Event Rate Per Participant Year During Study Period
Description: Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Severe and/or confirmed hypoglycemia event was a severe event or an event confirmed with plasma glucose =<70 mg/dL (=<3.9 mmol/L), or < 54 mg/dL (<3.0 mmol/L).
Time Frame: Day 1-Week 12, Week 13-Week 24, and 24 Week Period
Population: Safety population
Measure: Number; unit: Events per participant year
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
Events per participant year
  Any hypo Day1-Week12 | 8.93 | 11.31
  Any hypo Week13-14 | 11.28 | 11.60
  Any hypo 24 Week period | 10.09 | 11.45
  Severe and/or confirmed hypo (=<70mg/dL) D1-W12 | 8.08 | 10.47
  Severe and/or confirmed hypo (=<70mg/dL) W13-14 | 10.64 | 11.21
  Severe and/or confirmed hypo (≤70mg/dL) 24W period | 9.34 | 10.83
  Severe and/or confirmed hypo (< 54mg/dL) D1-W12 | 0.49 | 0.86
  Severe and/or confirmed hypo( <54 mg/dL) W13-14 | 0.73 | 0.91
  Severe and/or confirmed hypo (<54mg/dL) 24W period | 0.61 | 0.88

18. Other Pre Specified Outcome: Change From Baseline in Total Diabetes Treatment Satisfaction Questionnaire (DTSQ) Status at Week 12 and Week 24
Description: The DTSQs is a validated questionnaire to assess participant's satisfaction with their diabetes treatment. It consists of 8 items that are answered on a Likert scale from 0 to 6. Total treatment satisfaction score is the sum of items 1, 4-8 scores and ranged from 0 (no satisfaction) to 36 (high satisfaction with treatment). Adjusted least square means and standard errors were obtained from a mixed-effect model with MMRM.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT population. Number Analyzed = participants with at least one baseline and one post-baseline DTSQ status (DTSQs) total score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
score on a scale
  Week 12: number analyzed (Participants) | 438 | 436
  Week 12 | 5.08 (0.246) | 5.32 (0.245)
  Week 24: number analyzed (Participants) | 419 | 416
  Week 24 | 5.77 (0.257) | 5.44 (0.256)

19. Secondary Outcome: Hypoglycemia (Any, Severe and/or Confirmed Hypoglycemia: Nocturnal ) Event Rate Per Participant Year During Study Period
Description: Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Severe and/or confirmed hypoglycemia event was a severe event or an event confirmed with plasma glucose =<70 mg/dL (=<3.9 mmol/L), or < 54 mg/dL (<3.0 mmol/L). Nocturnal hypoglycemia was hypoglycemia that occurred between 00:00 and 05:59 hours (clock time).
Time Frame: Day 1-Week 12, Week 13-Week 24, and 24 Week Period
Population: Safety population
Measure: Number; unit: Events per participant year
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 462 | 462
Events per participant year
  Any hypo D1-W12 | 1.65 | 2.36
  Any hypo W13-14 | 2.32 | 2.39
  Any hypo 24Week period | 1.98 | 2.38
  Severe and/or confirmed hypo(=<70mg/dL)D1-W12 | 1.42 | 2.20
  Severe and/or confirmed hypo(=<70mg/dL)W13-14 | 2.24 | 2.33
  Severe and/or confirmed hypo(=<70mg/dL)24W Period | 1.83 | 2.26
  Severe and/or confirmed hypo(< 54mg/dL)D1-W12 | 0.16 | 0.19
  Severe and/or confirmed hypo(< 54mg/dL)W13-14 | 0.33 | 0.26
  Severe and/or confirmed hypo(< 54mg/dL)24W Period | 0.24 | 0.22

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected from signature of the informed consent form until 7 days after last treatment administration (maximum exposure: 24 Weeks).
Description: Reported adverse events and death were treatment-emergent adverse events that is adverse events that developed/worsened during the 'on treatment period' (On-treatment period was defined as the time from the first injection of open-label Investigational Medicinal Product (IMP) up to 7 days after the last injection of open-label IMP, regardless of the introduction of rescue therapy). Analysis was performed on safety population.
Arm/Group | Toujeo | Tresiba
All-Cause Mortality (participants affected / at risk) | 1/462 | 0/462
Serious Adverse Events (participants affected / at risk) | 21/462 | 20/462
Other Adverse Events (participants affected / at risk) | 56/462 | 58/462
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toujeo (N=462) | Tresiba (N=462)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 3 (3)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Artery Insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Retinal Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acoustic Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid Tumour Pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 3 (3)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Drug Use Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aortic Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0)
Varicose Ulceration (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toujeo (N=462) | Tresiba (N=462)
Upper Respiratory Tract Infection (Infections and infestations) | 24 (25) | 19 (20)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 38 (49) | 40 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2015-12-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT02738151/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT02738151/SAP_001.pdf